CLINICAL TRIAL: NCT03335709
Title: Evaluation of the Occupational Therapy Intervention Program "A Better Everyday Life 1.0" - a Protocol for a Feasibility Study
Brief Title: A Better Everyday Life 1.0 - a Protocol for a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Collaborators: University College of Northern Denmark (Other); University of Southern Denmark (Other); Municipality of Mariagerfjord, Denmark (Unknown)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, OT, PhD and senior researcher, Parker Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EW1
Record Dates: First submitted 2017-09-19; First posted 2017-11-08 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Activities of Daily Living
Keywords: Occupational therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADL intervention (Experimental): The participants are assigned to an eight-week intervention program aiming at enhancing ADL ability. The program consists of a minimum of five and a maximum of eight sessions; Session one - First meeting and occupational therapy evaluation (mandatory), Session two - Goal setting and clarifying reasons for problems related to ADL (mandatory), Session three- seven - Interventions aiming at enhancing ADL ability (Number of sessions can vary. However, a minimum of two sessions are mandatory), Session eight - Re-evaluation (Mandatory)
  Interventions: Behavioral: ADL intervention

INTERVENTIONS:
Behavioral: ADL intervention — Overall, an adaptational approach is being applied. The intervention sessions include changes related to the person, the environment and/or the occupation.

SUMMARY:
The purpose of the study is to evaluate a) the feasibility and b) the potential outcomes of a first version of an occupational therapy intervention program aiming at enhancing the ability to perform activities of daily living (ADL) among persons living with chronic conditions.

In the study a pre-post test design is applied.

DETAILED DESCRIPTION:
Introduction

Existing research has revealed that persons with chronic conditions experience decreased ability to perform both Personal ADL (PADL) and Instrumental ADL (IADL) tasks. Persons living with a chronic condition are offered various interventions. Besides medical treatment provided by physicians, to prevent or treat symptoms, persons with chronic diseases are often offered physical exercise in order to improve physical and/or mental body functions. Such interventions are founded on a belief that enhanced physical and mental body functioning also will result in improved ability to perform ADL tasks. However, existing research indicate that improvements in body functions not necessarily translate into improved ADL ability.

Research investigating the outcomes of rehabilitation services designed to enhance occupational performance, including ADL task performance, is sparse and insufficient. Existing research within this area is characterized by diversity and methodological limitations preventing development of clear intervention guidelines for clinical practice. Therefore, an occupational therapy program directly aiming at enhancing the ADL ability in persons with chronic conditions.

Aim

The purpose of this study is to evaluate a) the feasibility and b) the potential outcomes of a first version of an occupational therapy intervention program aiming at enhancing the ability to perform activities of daily living (ADL) among persons living with chronic conditions.

Methods

In the study a pre-test - post-test design is applied. That is, 30 participants living with chronic conditions are assigned to an eight week occupational therapy intervention program.

Outcome measures are self-reported and observed ADL ability measured using the ADL-Interview (ADL-I) and the Assessment of Motor and Process Skills (AMPS). Furthermore, various registrations (made by occupational therapists and participants) related to the feasibility of the intervention will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* diagnosed (by a physician) with one or more chronic condition(s)
* has participated in one or more the rehabilitation program at the municipality
* is living at home
* is experiencing problems related to performance of ADL tasks and is motivated to participate in the ADL intervention .

Exclusion Criteria:

* substance abuse
* other acute diagnoses affecting ADL task performance
* language barriers causing problems related to understanding Danish or participating in the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS) | Change from baseline at eight weeks.
  The Assessment of Motor and Process Skills (AMPS) is a standardized observation-based evaluation tool used by occupational therapists to measure a person's observed quality of ADL task performance in terms of physical effort and/or fatigue, efficiency, safety and independence. After the observation the quality of each skill is evaluated on a four point ordinal scale according to the scoring criteria in the AMPS manual.
  The available AMPS software, based on Many-Faceted Rasch statistics, makes it possible to convert ordinal raw scores into overall linear ADL motor and ADL process ability measures adjusted for task challenge, skill item difficulty and rater severity. The measures are expressed in logits (log-odds probability units).
ADL-Interview (ADL-I) | Change from baseline at eight weeks.
  The ADL-Interview (ADL-I) is developed to describe and measure the ADL ability based on self-report. Using the ADL-I, the participant is asked to report their perceived ADL ability (i.e. quality of ADL task performance) for each of the 47 ADL items using seven response categories.
  Data will be used to (a) describe the self-reported quality of ADL task performance on each task for a single person or a group of people and (b) measure a single person's overall self-reported quality of ADL task performance. To create an overall measure of self-reported quality of ADL task performance Rasch measurement methods are applied in order to transform the ratings into an overall linear (interval scale) measure of self-reported quality of ADL task performance, adjusted for the difficulty of the ADL task.

CONTACTS AND LOCATIONS:
Overall Officials: Eva E Wæhrens, PhD, Principal Investigator — The Parker Institute
Locations (1):
- Municipality of Mariagerfjord, Hadsund, Denmark

REFERENCES:
- [Derived] Nielsen KT, Guidetti S, von Bulow C, Klokker L, Waehrens EE. Feasibility of ABLE 1.0-a program aiming at enhancing the ability to perform activities of daily living in persons with chronic conditions. Pilot Feasibility Stud. 2021 Feb 18;7(1):52. doi: 10.1186/s40814-021-00790-7. PMID 33602338
- [Derived] Guidetti S, Nielsen KT, von Bulow C, Pilegaard MS, Klokker L, Waehrens EE. Evaluation of an intervention programme addressing ability to perform activities of daily living among persons with chronic conditions: study protocol for a feasibility trial (ABLE). BMJ Open. 2018 May 20;8(5):e020812. doi: 10.1136/bmjopen-2017-020812. PMID 29780029